CLINICAL TRIAL: NCT02808260
Title: Predicting Development of Sub-Clinical Atrial Fibrillation in Device Patients
Brief Title: Predicting Development of SCAF in Device Patients
Status: Recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Genome Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 20160338
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
Keywords: sub-clinical atrial fibrillation; biomarkers; implanted pacemaker or defibrillator
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for the measurement of biomarkers
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Atrial fibrillation (AF) often starts with short episodes of rapid irregular heartbeats that are only detected by implanted pacemakers or defibrillators. Usually people don't know that they have these episodes. Over time, these episodes can happen more often and last for longer periods. In some people, the heart eventually remains permanently in a fast irregular rhythm, known as atrial fibrillation. This condition can lead to strokes and blood clots. If physicians could detect atrial fibrillation at a very early stage they could treat people early and possibly prevent the condition from becoming permanent. People with implanted devices allow a unique opportunity to constantly monitor the heart rhythm so investigators can detect any irregularities immediately.

Investigators don't know which people are at risk of developing short episodes of fast irregular heartbeats that can lead to atrial fibrillation. The purpose of this study is to find out if there are proteins or chemical changes in the blood that can predict the risk of developing atrial fibrillation. These chemical changes, also known as biomarkers, may also be able to give investigators other clues about atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is considered to be a progressive condition that starts with episodes of paroxysmal AF (short runs of AF), progresses to persistent AF (can be reverted to normal rhythm) and eventually to permanent AF. More than 25% of people with paroxysmal AF will go on to develop persistent or chronic atrial fibrillation. The progression rate is around 5% per annum. AF can result in devastating outcomes such as stroke/TIA and systemic embolic events. In people with implanted devices such as ICDs, investigators can detect non-symptomatic rapid atrial arrhythmia, known as subclinical atrial fibrillation (SCAF), before it becomes symptomatic. In the ASSERT trial, SCAF was detected in 10% of patients with newly implanted devices within the first 3 months. Of these, nearly 16% developed clinical atrial fibrillation within 2.5 years vs 3% in those who did not exhibit SCAF within the first 3 months. During the follow up period, a further 24.5% of patients developed SCAF. People with SCAF also had a higher risk of stroke and systemic embolism.

Earlier diagnosis and treatment of AF may lead to better prevention and outcomes. The availability of serum based biomarkers that can predict the early onset of atrial fibrillation, may help in the identification of patients at risk for developing AF early. This would also allow the identification of the patient population most suitable for the evaluation of possible future intervention strategies to prevent the onset of atrial fibrillation, and alter its natural history and complications.

In this study investigators will study patients that have a permanent pacemaker or defibrillator implanted. These devices continuously monitor the patient's heart rhythm, detecting any irregularities. Patients with these devices are followed up in outpatient clinics on a regular basis. The information from the devices is downloaded at each follow up visit and analyzed by staff in the clinic.

Investigators will recruit patients for this study after the device was implanted. After obtaining consent, investigators will collect a blood sample for measuring biomarkers. They will interview the participant in regards to previous health history, smoking, alcohol consumption, family history and current medications. Participants' medical records will be reviewed annually for the next 10 years, to monitor for any irregular heart rhythms, hospitalizations and death.

ELIGIBILITY:
Inclusion Criteria:

• Dual chamber permanent pacemaker or defibrillator implanted within previous 10 years

Exclusion Criteria:

* Clinical atrial fibrillation documented by surface ECG (12 lead ECG, Telemetry, Holter)
* Participants considered by the investigator to be unsuitable for the study for the following reason: life expectancy less than 2 years due to concomitant disease
* Participants who are pregnant or breast-feeding
* Congenital heart disease
* Inherited arrhythmia syndrome, i.e. Brugada, long QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will recruit patients with a permanent defibrillator or pacemaker who have an upcoming appointment at the Device Clinic.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
The development of new Sub-Clinical Atrial Fibrillation as recorded on implanted devices | 11 years
  Participants will be monitored by clinical follow up for a year and then medical record reviews for an additional 10 years
Sub-clinical Atrial Fibrillation as predicted by biomarkers | 11 years
  Biomarkers will be measured at baseline and after 1 year to see if biomarkers can predict which people will develop sub-clinical atrial fibrillation during the 11 year follow up period

SECONDARY OUTCOMES:
The development of clinical atrial fibrillation, including persistent atrial fibrillation. | 11 years
  The investigators will monitor participants to see how many develop persistent atrial fibrillation within 11 years of device implant

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Nery, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No